CLINICAL TRIAL: NCT06993467
Title: Oxygen Delivery During Cardiopulmonary Bypass And Inflammatory Reaction After Cardiac Surgery
Acronym: OXYINFLAMM
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Enrico Squiccimarro, Dr, Azienda Ospedaliero, Universitaria Ospedali Riuniti
Other Study IDs: OXY_INFLAMM.01
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery; Systemic Inflammatory Response Syndrome (SIRS)
Keywords: cardiopulmonary bypass; oxygen delivery; systemic inflammatory reaction syndrome; cardiac surgery
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac surgery, especially when involving cardiopulmonary bypass (CPB), has long been associated with a systemic inflammatory response that can lead to a range of complications, from mild symptoms to severe organ dysfunction, and mortality. The exact mechanisms behind this response remain a topic of extensive research, but it's clear that the body's reaction to the extracorporeal circulation, combined with surgical trauma, plays a significant role. Factors such as genomics, age, specific preoperative conditions, and the duration of operations have been associated with significant clinical responses.

A pivotal insight into this response comes from recent genome-wide transcriptional analyses. Perioperative ischemia and ischemia-reperfusion injury (IRI) have been suggested as hub-nodes in a hierarchic structure evaluating the response to cardiac surgery. This suggests that IRI isn't just a side effect of the surgery but might be a central player in the body's inflammatory response. The role of perioperative ischemia and its potential as a significant contributor to the postoperative inflammatory response cannot be understated. This study aims to delve deeper into the role of oxygen delivery and its implications in the systemic inflammatory response post- cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-90 years)
* Elective surgery
* CPB-assisted

Exclusion Criteria:

* Age < 18 or > 90 years
* Infective endocarditis
* Hypothermia during surgery (<34°C)
* Emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients undergoing elective cardiopulmonary bypass-assisted procedures
Sampling Method: Probability Sample
Enrollment: 908 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
SIRS | 12 hours after surgery
  Systemic Inflammatory Reaction Syndrome (SIRS) as per the 1991 American College of Chest Physicians/Society of Critical Care Medicine criteria

SECONDARY OUTCOMES:
Composite outcome | Up to 30 days
  Composite outcome comprising death, TIA/stroke, renal replacement therapy, bleeding, mechanical circulatory support, or ICU stay >96 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Anthea Hospital, Bari, Italia
  - Santa Maria Hospital, GVM Care & Research, Bari, Italia

IPD SHARING:
Plan to Share IPD: Undecided